CLINICAL TRIAL: NCT02350738
Title: Effects of Multimodal Cognitive Enhancement Therapy (MCET) for People With Mild Cognitive Impairment and Early Stage Dementia: a Randomized, Controlled, Double-blind, Cross-over Trial
Brief Title: Effects of Multimodal Cognitive Enhancement Therapy (MCET) for Ealy Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ki Woong Kim (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Ki Woong Kim, Professor, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SeoulNUBH
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Mild Cognitive Impairment; Dementia, Mild
Keywords: Mild cognitive impairment; Dementia; Cognitive training; Cognitive rehabilitation; Cognitive therapy
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCET_Mock group (Experimental): Period I: MCET for 8 weeks (3 sessions/ week); Washout for 4 weeks and cross-over; Period II: mock therapy for 8 weeks (3 sessions/week)
  Interventions: Other: Period I MCET (8 wks); Other: Washout (4 wks)
- Mock_MCET group (Experimental): Period I: mock therapy for 8 weeks (3 sessions/week); Washout for 4 weeks cross-over; Period II: MCET for 8 weeks (3 sessions/ week);
  Interventions: Other: Washout (4 wks); Other: Period II MCET (8 wks)

INTERVENTIONS:
Other: Period I MCET (8 wks) — MCET_Mock group: Multimodal Cognitive Enhancement Therapy (MCET) (3 sessions/wk) Mock_MCET group: mock-therapy (3 sessions/wk)
  Arms: MCET_Mock group
Other: Washout (4 wks) — 4 weeks wash-out period in both arms and cross-over
Other: Period II MCET (8 wks) — MCET_Mock group: mock therapy (MCET) (3 sessions/wk) Mock_MCET group: Multimodal Cognitive Enhancement Therapy (MCET) (3 sessions/wk)
  Arms: Mock_MCET group

SUMMARY:
This study evaluates the effects of Multimodal Cognitive Enhancement Therapy (MCET) for people with mild cognitive impairment and early stage dementia by a randomized, controlled (mock-therapy), double-blind, cross-over trial

DETAILED DESCRIPTION:
Multimodal Cognitive Enhancement Therapy (MCET) was developed for cognitive rehabilitation of mild cognitive impairment or ealy dementia. MCET consists of cognitive training, cognitive stimulation, reality orientation, physical therapy, reminiscence therapy and music therapy that obtained 'A' grade of recommendation by SIGN(Scottish Intercollegiate Guidelines Network) for their efficacy (one of the followings: global cognition/specific cognitive domain/mood/activities of daily living/behavioral and psychological symptoms/quality of life) based on the systematic review and meta-analysis performed by our research team.

This study investigated the efficacy of MCET compared with mock-therapy that consisted of random activities that were not based on clinical evidences (e.g., watching TV, conversation etc.).

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-90
* Diagnosed to dementia by the Diagnostic and Statistical Manual, fourth edition (DSM-IV) or to mild cognitive impairment by International Working Group on Mild Cognitive Impairment
* Clinical Dementia Rating (CDR) of 0 or 0.5 for mild cognitive impairment, 0.5 or 1 for early dementia

Exclusion Criteria:

* Evidence of current delirium, confusion
* Any acute neurological conditions (infectious or inflammatory disorders such as viral, fungal or syphilis) or acute medical conditions
* Current major psychiatric disorder by DSM-IV such as major depressive episode or manic or psychotic episode

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in the Mini-Mental State Examination for dementia screening before and after period I and before and after period II intervention (crossover part of the study) | baseline, week8 (after period 1), week 20 (after period 2), 6 months after period 2
  To evaluate the effect on the global cognition

SECONDARY OUTCOMES:
Change in the Korean version of Alzheimer's Disease Assessment Scale -cognitive subscale of Korean version (ADAS-KCog) before and after period I and before and after period II intervention (crossover part of the study) | baseline, week8 (after period 1), week 20 (after period 2), 6 months after period 2
  To evaluate the effect on global cognition
Change in the Disability Assessment for Dementia (DAD-K) before and after period I and before and after period II intervention (crossover part of the study) | baseline, week8 (after period 1), week 20 (after period 2), 6 months after period 2
  To evaluate the effect on the functional level (basic/instrumental activities of daily living)
Change in the Revised Memory and Behavior Problems Checklist (RMBPC) before and after period I and before and after period II intervention (crossover part of the study) | baseline, week8 (after period 1), week 20 (after period 2), 6 months after period 2
  To evaluate the effect on the behavioral and psychological symptoms of dementia
Change in the Quality of Life-AD (QoL-AD) of patients before and after period I and before and after period II intervention (crossover part of the study) | baseline, week8 (after period 1), week 20 (after period 2), 6 months after period 2
  To evaluate the effect on the patient's self-rating quality of life
Change in the Quality of Life-AD (QoL-AD) of caregivers before and after period I and before and after period II intervention (crossover part of the study) | baseline, week8 (after period 1), week 20 (after period 2), 6 months after period 2
  To evaluate the effect on the patient's quality of life evaluated by his/her caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea